CLINICAL TRIAL: NCT04745572
Title: Development of an Adaptive Treatment Strategy for Weight Loss in People With Prediabetes Using a Sequential Multiple Assignment Randomized Trial
Brief Title: Development of an Adaptive Treatment for Weight Loss in People With Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: General Mills (Industry)
Responsible Party: Principal Investigator, Holly Wyatt, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300006816; General Mills (Other Grant/Funding Number: General Mills)
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2024-10

CONDITIONS: PreDiabetes; Obesity
Keywords: weight loss; reduced carbohydrate diet; exercise training; time restricted eating
MeSH Terms: conditions — Prediabetic State; Obesity; Weight Loss; Intermittent Fasting | interventions — Diet, High-Protein Low-Carbohydrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Carbohydrate Diet (Experimental): Enrollment in a group-based behavioral weight loss intervention based on the Diabetes Prevention Program curriculum with high carbohydrate diet plan.
  Interventions: Behavioral: High Carbohydrate Diet
- Reduced Carbohydrate Diet (Experimental): Enrollment in a group-based behavioral weight loss intervention based on the Diabetes Prevention Program curriculum with reduced carbohydrate diet plan.
  Interventions: Behavioral: Reduced Carbohydrate Diet

INTERVENTIONS:
Behavioral: High Carbohydrate Diet — Participants randomized to this group will participate in a group-based weight behavioral management program and consume a high carbohydrate (HC) diet. Because this protocol uses a sequential, multiple assignment, randomized trial (SMART) design, response will be assessed at week 4. Responders will continue with their 1st stage assignment for the remainder of the study. Non-responders will be randomized to 2nd stage intervention of either combine HC diet with time-restricted eating (TRE) or HC diet with additional exercise counseling and support.
  Arms: High Carbohydrate Diet
Behavioral: Reduced Carbohydrate Diet — Participants randomized to this group will participate in a group-based behavioral weight management program and consume a reduced carbohydrate (RC) diet. Because this is a sequential, multiple assignment, randomized trial (SMART) design, response will be assessed at week 4. Responders will continue with their 1st stage assignment for the remainder of the study. Non-responders will be randomized to 2nd stage intervention of either combine RC diet with time-restricted eating (TRE) or RC diet with additional exercise counseling and support.
  Arms: Reduced Carbohydrate Diet

SUMMARY:
This 16-week study will use an experimental approach called the Sequential Multiple Assignment Randomized Trial to help determine which combination and sequence of weight loss program features are most effective in people who are at risk for type 2 diabetes. Participants in the study will be initially randomized to consume either a high or reduced carbohydrate diet. After 4 weeks, participants will be identified as Responders (greater than or equal to 2.5% weight loss) or Non-Responders (less than 2.5% weight loss). Responders will continue with their initial randomized group for the remainder of the trial. Non-responders will be re-randomized to 2nd stage interventions of either including additional exercise counseling and training or beginning a time restricted eating protocol for the remainder of the trial.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* BMI of 27 kg/m2 or greater
* at risk for developing type 2 diabetes (prediabetes)

Exclusion Criteria:

* Pregnant, planning to become pregnant, or breastfeeding
* uncontrolled hypo or hyperthyroidism

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Changes in body weight | week 16 visit
  Measured on digital scale at final visit.

SECONDARY OUTCOMES:
Change in glucose | week 16 visit
  Serum glucose will be measured in a fasted state.
Change in hemoglobin A1c | week 16 visit
  A1c is a measure of average glucose over the previous 3 months.
Change in insulin | week 16 visit
  Serum insulin will be measured in a fasted state.
Changes in QUICKI index | week 16 visit
  Predictor of insulin resistance that will be calculated from glucose and insulin measures

OTHER OUTCOMES:
Changes in fat mass | week 16 visit
  As measured by bioelectrical impedance analysis (BIA) on the InBody S10 body composition analyzer.
Changes in lipids | week 16 visit
  Fasting serum concentrations of total cholesterol, HDL cholesterol, triglycerides, and LDL cholesterol
Change in Blood Pressure | week 16 visit
  Measured with a clinical grade blood pressure cuff.
Changes in body weight | week 4 visit
  Measured on digital scale in order to determine "responder" or "non-responder" status.
Changes in aerobic fitness | week 16 visit
  As measured by the 3-minute step test.
Changes in overall strength | week 16 visit
  As measured by hand grip dynamometry
Diet Intake and Physical Activity Monitoring | week 16 visit
  7-day food logs and weekly physical activity logs
Diet Intake and Physical Activity Monitoring | week 4 visit
  7-day food logs and weekly physical activity logs

CONTACTS AND LOCATIONS:
Overall Officials: Holly Wyatt, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Highlands Family and Community Medicine Clinic, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ellison KM, El Zein A, Baidwan NK, Ferguson CC, Fowler LA, Bryan DR, Reynolds C, Hermanson D, Berg KJ, Mehta T, Hill JO, Wyatt HR, Sayer RD. Adaptive dietary and exercise strategies for weight loss in Adults with Prediabetes Trial (ADAPT): a sequential multiple assignment randomized trial. Am J Clin Nutr. 2025 Oct;122(4):1093-1102. doi: 10.1016/j.ajcnut.2025.07.034. Epub 2025 Aug 7. PMID 40763896